CLINICAL TRIAL: NCT06334341
Title: A Multilevel, Multiphase Optimization Strategy for PrEP: Patients and Providers in Primary Care
Brief Title: A Multilevel, Multiphase Optimization Strategy for PrEP (MOST:PrEP)
Acronym: MOST:PrEP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of South Florida (Other); New York University (Other)
Responsible Party: Principal Investigator, Elizabeth Lockhart, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: R01MD018523-01A1 (NIH)
Record Dates: First submitted 2024-03-18; First posted 2024-03-28 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: HIV Seropositivity
Keywords: Preexposure Prophylaxis
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- No intervention (No Intervention): No intervention
- Video (Experimental): Patient PrEP Video only
  Interventions: Behavioral: PrEP Informational Video
- Risk Assessment (Experimental): Patient Risk Assessment only
  Interventions: Behavioral: HIV Risk Assessment
- Risk Assessment and Video (Experimental): Patient Risk Assessment and Patient PrEP Video
  Interventions: Behavioral: HIV Risk Assessment; Behavioral: PrEP Informational Video
- Best Practice Alert (Experimental): Best Practice Alert only
  Interventions: Behavioral: Best Practice Alert
- Best Practice Alert and Video (Experimental): Best Practice Alert and Patient PrEP Video
  Interventions: Behavioral: Best Practice Alert; Behavioral: PrEP Informational Video
- Best Practice Alert and Risk Assessment (Experimental): Best Practice Alert and Patient Risk Assessment
  Interventions: Behavioral: Best Practice Alert
- Best Practice Alert, Risk Assessment and Video (Experimental): Best Practice Alert, Patient Risk Assessment, and Patient PrEP Video
  Interventions: Behavioral: Best Practice Alert; Behavioral: HIV Risk Assessment; Behavioral: PrEP Informational Video
- Training (Experimental): Provider Training
  Interventions: Behavioral: Computer-based simulation training for providers
- Training and Video (Experimental): Provider Training and Patient PrEP Video
  Interventions: Behavioral: Computer-based simulation training for providers; Behavioral: PrEP Informational Video
- Training and Risk Assessment (Experimental): Provider Training and Patient Risk Assessment
  Interventions: Behavioral: Computer-based simulation training for providers; Behavioral: HIV Risk Assessment
- Training, Risk Assessment, and Video (Experimental): Provider Training, Patient Risk Assessment, and Patient PrEP Video
  Interventions: Behavioral: Computer-based simulation training for providers; Behavioral: HIV Risk Assessment; Behavioral: PrEP Informational Video
- Training and Best Practice Alert (Experimental): Provider Training and Best Practice Alert
  Interventions: Behavioral: Computer-based simulation training for providers; Behavioral: Best Practice Alert
- Training, Best Practice Alert, and Video (Experimental): Provider Training, Best Practice Alert, and Patient PrEP Video
  Interventions: Behavioral: Computer-based simulation training for providers; Behavioral: Best Practice Alert; Behavioral: PrEP Informational Video
- Training, Best Practice Alert, and Risk Assessment (Experimental): Provider Training, Best Practice Alert, and Patient Risk Assessment
  Interventions: Behavioral: Computer-based simulation training for providers; Behavioral: Best Practice Alert; Behavioral: HIV Risk Assessment
- Training, Best Practice Alert, Risk Assessment, and Video (Experimental): Provider Training, Best Practice Alert, Patient Risk Assessment, and Patient PrEP Video
  Interventions: Behavioral: Computer-based simulation training for providers; Behavioral: Best Practice Alert; Behavioral: HIV Risk Assessment; Behavioral: PrEP Informational Video

INTERVENTIONS:
Behavioral: Computer-based simulation training for providers — A Computer-Based Simulation training for providers, based on the Centers for Disease Control and Prevention "Guide for Healthcare Professional: Discussing Sexual Health with Your Patients", current PrEP information, and the Social Cognitive Theory. This is a single-session, 30-minute training module contains educational information with animated narration about PrEP, how to take a sexual health history, understanding internal bias, potential patient barriers to PrEP as well as recorded video-simulated encounters, in which providers view different types of patient/provider interactions.
  Arms: Training; Training and Best Practice Alert; Training and Risk Assessment; Training and Video; Training, Best Practice Alert, Risk Assessment, and Video; Training, Best Practice Alert, and Risk Assessment; Training, Best Practice Alert, and Video; Training, Risk Assessment, and Video
Behavioral: Best Practice Alert — A Best Practice Alert will alert providers to patients who are part of the Centers for Disease Control and Prevention PrEP priority populations.
  Arms: Best Practice Alert; Best Practice Alert and Risk Assessment; Best Practice Alert and Video; Best Practice Alert, Risk Assessment and Video; Training and Best Practice Alert; Training, Best Practice Alert, Risk Assessment, and Video; Training, Best Practice Alert, and Risk Assessment; Training, Best Practice Alert, and Video
Behavioral: HIV Risk Assessment — A risk assessment tool that considers the behaviors - i.e., types of sexual activities, protective behaviors (condoms, PrEP, ART), and other factors (HIV status, sexually transmitted infections) of the respondent.
  Arms: Best Practice Alert, Risk Assessment and Video; Risk Assessment; Risk Assessment and Video; Training and Risk Assessment; Training, Best Practice Alert, Risk Assessment, and Video; Training, Best Practice Alert, and Risk Assessment; Training, Risk Assessment, and Video
Behavioral: PrEP Informational Video — A short informational video, tailored to the local Detroit context with themes that will focus on introducing PrEP, stigma surrounding taking PrEP, and potential barriers and how to overcome them.
  Arms: Best Practice Alert and Video; Best Practice Alert, Risk Assessment and Video; Risk Assessment and Video; Training and Video; Training, Best Practice Alert, Risk Assessment, and Video; Training, Best Practice Alert, and Video; Training, Risk Assessment, and Video; Video

SUMMARY:
What is known: There are 1.2 million people in the US who meet the indications for PrEP; yet, disparities exist in uptake. For example, only 9% of Black and 16% of Latino individuals, compared to 65% of White individuals, have been prescribed PrEP. At Henry Ford Health (HFH) system, only 10% of eligible patients have been prescribed PrEP. Primary care is an ideal setting for PrEP to be offered as an HIV prevention method since providers see large numbers of patients who are HIV negative, with some who are at increased risk for HIV, and the primary care setting is often the point of entry to the healthcare system. The multiphase optimization strategy (MOST) framework is a novel, innovative way to identify an efficient intervention. What will be done: In this optimization trial, the investigators will test the effectiveness of intervention components, alone and in combination, on new PrEP prescriptions in primary care at HFH. First, feedback will be generated on context-specific (system and individual level) factors for intervention component delivery via focus groups with providers (n=15) and patients eligible for PrEP (n=30). Then, four intervention components will be tested in an optimization trial, with 16 conditions being implemented at 32 clinics. Finally, feedback will be generated on the factors that affected implementation via semi-structured interviews with providers (n=30) and patients (n=30). Participants will be primary care providers (PCPs) and patients eligible for PrEP in Henry Ford Health System. Clinics will be randomized (yes/no) to receive any combination of provider and patient intervention components. Provider intervention components include computer-based simulation training and/or best practice alerts delivered via the electronic health record (EHR). Patient intervention components include HIV risk assessment and/or PrEP informational video - both delivered via the EHR. Primary outcome is the rate of new PrEP prescriptions at the clinic level. Secondary outcomes will include PrEP maintenance, number of HIV tests ordered by a PCP, and number of PCPs trained. Sub analyses will test which factors moderate (e.g., patient sex, race, age, gender, sexual orientation) or mediate (e.g., perceived HIV risk, provider and patient PrEP knowledge) PrEP uptake, focusing on priority populations and disparities in rates of PrEP prescription. Implications: 1) Understanding which intervention components lead to increased PrEP prescriptions will represent an important advance in HIV prevention efforts. 2) Optimizing a multi-level intervention for providers and patients to increase PrEP prescriptions would lead to a new, efficient, evidence-based option. 3) Determining what factors are related to PrEP uptake will help reduce disparities in PrEP initiation among those most in need. 4) Understanding the context specific factors related to intervention component implementation will help identify best methods for replication/adaptation in other healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Provider:≥ 18-years old
* Provider: employed at HFH as a primary care provider
* Provider: eligible to write prescriptions in the state of Michigan
* Patient: ≥ 18 years old
* Patient: have an appointment with a Henry Ford primary care clinic during the study period
* Patient: have an EHR account
* Patient: meet the indications for PrEP

Exclusion Criteria:

* Provider: not a HFH primary care provider
* Provider: does not have prescribing privileges in the state of Michigan
* Patient: currently prescribed or taking PrEP
* Patient: living with HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Clinic-Level PrEP Prescription | Year 1 and Year 5 electronic health record data pull.
  The number of new PrEP prescriptions written within 6-months of the study-associated patient appointment. It is defined as a new documented prescription in the patient electronic health records for PrEP (daily pill or injection) at any date between the initial study primary care appointment plus 180 days.

SECONDARY OUTCOMES:
PrEP Knowledge | Provider pre-post survey and patient demographic and 6- month surveys
  PrEP knowledge will be measured by 6-items assessing PrEP dosing frequency, approved FDA medications, HIV antibody testing prior to PrEP initiation, HIV testing frequency while on PrEP, contraindications to prescribing PrEP, and routine standard of care practices for patients taking PrEP
PrEP awareness | Provider pre-post survey and patient demographic and 6- month surveys
  PrEP awareness will be measured by the statement "there is a pill (drug/medication) that a person can take to prevent transmission of HIV from an infected (HIV positive) sex partner to an uninfected (HIV negative) partner." with responses true/false, don't know.
PrEP prescribing comfort | Pre-intervention and immediately after the intervention for providers
  PrEP prescribing comfort will be measured by 9- items from the PrEP Information, Motivation, and Behaviors survey.
PrEP prescribing intentions | Pre-intervention and immediately after the intervention for providers
  PrEP prescribing intentions will be measured by 8- items from the PrEP Information, Motivation, and Behaviors survey.
Perceived HIV risk | Patient demographic and 6- month surveys
  Patients perceived HIV risk will be measured by 10- items from the Perceived Risk of HIV scale.
Preferences for patient- provider communication | Patient demographic and 6- month surveys
  Preferences for patient-provider communications will be measured by the Control Preferences Scale, the Communication Assessment Tool, and the Patient-Practitioner Orientation Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Lockhart, PhD, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No